CLINICAL TRIAL: NCT01183871
Title: Changes in Cerebral Oxygenation in Patients With Pulmonary Dysfunction After Lung Resection
Brief Title: Cerebral Oxygenation After Lung Resection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King Faisal University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 201011
Record Dates: First submitted 2010-08-12; First posted 2010-08-18 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Elective; Lung Resection; Surgery
Keywords: Cerebral oxygenation; thoracotomy; lung resection; pulmonary dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- good pulmonary functions (group 1) (Active Comparator): FVC and/or FEV1 of 80% of predicted or more
  Interventions: Procedure: Monitoring of cerebral oxygenation
- mild pulmonary dysfunction (group 2) (Active Comparator): FVC and/or FEV1 of 70%-79% of predicted
  Interventions: Procedure: Monitoring of cerebral oxygenation
- moderate pulmonary dysfunction (group 3) (Active Comparator): FVC and/or FEV1 of 60%-69% of predicted
  Interventions: Procedure: Monitoring of cerebral oxygenation
- severe pulmonary dysfunction (group 4) (Active Comparator): FVC and/or FEV1 of 50%-59% of predicted
  Interventions: Procedure: Monitoring of cerebral oxygenation

INTERVENTIONS:
Procedure: Monitoring of cerebral oxygenation — The internal jugular vein will be cannulated using ultrasound guidance in a cephalad direction, using the Seldinger J-shaped guidewire and it will be advanced only for 2-3 cm beyond the needle insertion site to avoid vascular injury to the jugular bulb. At which point the catheter is advanced until resistance is met at the jugular bulb, usually about 15 cm. The catheter is then pulled back 0.5-1.0 cm so that the catheter does not continue to abut the roof of the jugular bulb and to minimize the cephalad vascular impact with head movement, thereby reducing the risk of vascular injury. Skull x-ray will be used to confirm placement.

SUMMARY:
The investigators hypothesize that the lung resection would be associated with lower jugular bulb oxygen saturation in patients with severe pulmonary dysfunction than in patients with healthy lung functions.

DETAILED DESCRIPTION:
Surgery remains the treatment of choice for patients with resectable lung cancer. However, a significant proportion of patients undergoing lung resections have the associated condition COPD,1 which increases the risk of perioperative complications and death. New techniques in anesthesiology and critical care have enabled patients with COPD to have better outcomes following lung resections. Nowadays, patients with limited lung function, who would have been denied surgery according to the criteria proposed in the past, may undergo pulmonary resection with a low mortality rate.2

Lung resection results in loss of lung parenchyma including residual healthy lung tissue and in reduction in the pulmonary vascular bed. A decrease in residual pulmonary vascular bed after lung resection causes an increase in the right heart afterload, and in others, it would be associated with an increase in the right heart preload.3

The removal of lung parenchyma from patients with carcinoma of the lung, may lead to cardiopulmonary failure or death. A predicted postoperative forced expiratory volume in one second (FEV1) less than 0.8 to 1.0 liter is considered an indicative of a high risk of postoperative chronic ventilatory insufficiency. After pneumonectomy, FEV1 decreases by 29-35% and forced vital capacity (FVC) decreases by 27-44%. After lobectomy, FEV1 and FVC decrease to12-23% and 10-30%, respectively.4

After lobectomy in patients with normal pulmonary functions, there is a transient good maintenance of gas exchange for only 6-12hours, then it is followed with progressive deterioration in oxygen delivery and intra-pulmonary shunt fraction because of peripheral atelectasis 4-13 days after surgery.5 Other investigators reported a significant decrease in maximal oxygen uptake (VO2-Max) and maximal work rate (WR-Max) by 27% and 42%, respectively, 3 months after pneumonectomy, and by13% and 2%, respectively after lobectomy.

In patients with moderate-to-severe pulmonary dysfunction there is significant worsening of pulmonary gas exchange; especially during one-lung ventilation (OLV) which is the mandatory technique to facilitate thoracic surgery. This worsening is more marked in patients undergoing right thoracotomies after lung resection.6

Postoperative lung function changes in the elderly followed the similar trend as in patients with pulmonary dysfunction. The mean postoperative decrease in FEV 1 was 14.16% in the elderly, compared with a 29.23% decrease in patients with normal lung function ( P < 0.05). However, the operative morbidity in the elderly group was significantly lower than in patients with pulmonary dysfunction (23.3% vs. 60%).7

The potential for postoperative neurocognitive dysfunction and its impact on the postoperative course has gained recent attention over the past few years.8 There is an interesting study for the changes in brain tissue oxygenation (rSO2) during OLV for thoracic surgery using near infrared spectroscopy (NIRS), otherwise known as cerebral oximetry, is a non-invasive device that uses infrared light to estimate brain tissue oxygenation which may occur during OLV. The investigators reported significant changes in rSO2 occur during OLV for thoracic surgical procedures without changes in hemodynamic or ventilatory parameters. They recommended future studies to determine the impact of such changes on the postoperative course of these patients.9

According to the above evidences, the changes in oxygen delivery, oxygen uptake and intrapulmonary shunt after lung resection will be reflected on the cerebral blood flow and oxygen delivery and jugular bulb oxygen saturation in patients with impaired pulmonary functions rather than those with healthy lung functions.

Oxygenation of cerebral venous outflow has been investigated as a neuro-monitor for more than 50 years.10-12 Currently, jugular venous oxygen saturation (SjVO2) provides an indirect assessment of cerebral oxygen use and is used to guide physiologic management decisions in a variety of clinical paradigms.13-14 This is simply can be achieved through introducing of an intravascular catheter, similar to those used for central venous pressure monitoring, may be placed retrograde, via the internal jugular vein, into the jugular bulb at the base of skull.15

Jugular venous oxygen is an indirect assessment of cerebral oxygen use. Simplistically, when demand exceeds supply, the brain extracts greater oxygen, resulting in decreased jugular bulb oxygen saturation. If cerebral blood flow (CBF) decreases, a point is eventually reached at which the brain can no longer completely compensate for decreased CBF by a further increase in oxygen extraction. At this point, oxygen consumption decreases and anaerobic metabolism with lactate production ensues. When cerebral oxygen supply exceeds demand, oxygen saturation of jugular bulb blood is increased.15

To our knowledge there is no any study was done on the changes in cerebral oxygenation after lung resections, especially in the high-risk group with pulmonary dysfunction.

Project Objectives:

We hypothesize that the lung resection would be associated with lower jugular bulb oxygen saturation in the patients with severe pulmonary dysfunction than in the patients with healthy lung functions.

ELIGIBILITY:
Inclusion Criteria:

* ASA II-IV
* Ages 18-60 yrs.
* Good or impaired pulmonary function tests

Exclusion Criteria:

* Decompensated cardiac function (>New York Heart Association II).
* Hepatic and renal diseases
* Arrhythmias
* Moderate pulmonary hypertension (mean pulmonary artery pressure (MPAP) >35 mm Hg),
* Previous history of pneumonectomy, bilobectomy or lobectomy
* Cervical spine injury
* Tracheostomy
* Coagulopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
jugular bulb oxygenation | before (baseline) and15 min after induction of anesthesia during two-lung ventilation, 15, 30, 60 min after OLV, and 15 min after resuming of two-lung ventilation (TLV), and 1, 4, 6, 12, 18 and 24 hrs after recovery.
  jugular bulb oxygen saturation (SjvO2), estimated cerebral metabolic rate of oxygen [CMRO2], cerebral extraction of oxygen [CEO2], cerebral blood flow equivalent [CBFE], and arterial to jugular difference in oxygen content (AjvDO2)

SECONDARY OUTCOMES:
Respiratory and Hemodynamic Data | baseline and15 min after induction of anesthesia during two-lung ventilation,1, 4, 6, 12, 18 and 24 hrs after recovery.
  arterial oxygen saturation (SaO2,) arterial oxygen and carbon dioxide tensions (PaO2, and PaCO2, respectively), FEV1 FVC, HR, MAP,

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, M.D., Study Director — King Faisal University
Locations (1):
- King Fahd hospital of the University of Dammam, Khobar, Eastern Province, Saudi Arabia